CLINICAL TRIAL: NCT01260818
Title: Prospective Randomized Trial Comparing Topical Tranexamic Acid Plus Standard Of Care Versus Standard Of Care For The Reduction Of Blood Loss Following Primary Total Hip Arthroplasty Surgery
Brief Title: Topical Application of Tranexamic Acid Reduces Postoperative Blood Loss in Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: the First Affiliated Hospital of Guangzhou TCM University, the First Affiliated Hospital of Guangzhou TCM University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GZTCM-201001
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2010-12

CONDITIONS: Hip Replacement; Postoperative Hemorrhage
Keywords: Tranexamic Acid
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (Experimental)
  Interventions: Drug: Tranexamic Acid
- control group (Placebo Comparator)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Tranexamic Acid — 1 g Tranexamic Acid mixed with 100ml saline are kept in wound for 2 hours before drainage is opened postoperatively
  Arms: Tranexamic Acid
Drug: normal saline — 100ml saline is kept in wound for 2 hours before drainage is opened postoperatively
  Arms: control group

SUMMARY:
Tranexamic acid has been shown to reduce postoperative blood losses and transfusion requirements in a number of types of surgery. Most trials in orthopedic surgery have been conducted intravenously in arthroplasty, hip fracture and spine surgeries. This study would aim to see the effect of topical use of tranexamic acid in reduction of blood loss and transfusions for total hip arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* Patient who are to undergo elective total hip arthroplasty.
* Must be primary arthroplasty.
* Must be single-side arthroplasty.
* Must be older than 18 years.

Exclusion Criteria:

* Cemented arthroplasty.
* Patients with a platelet count less than 100, 000/mm3 or history of thrombocytopenia .
* Patients with known coagulopathy (APTT or PT outside normal range pre-operatively).
* Patients who have a past medical history of thrombi-embolism at any time.
* Patients with anemia (hemoglobin levels less than 8 mg/dl or hematocrit <24%).
* Patients with documented DVT or PE at screening or in past three months.
* Patients having known hypersensitivity to tranexamic acid or any other. constituent of the product.
* Patients with any associated major illness (e.g., severe cardiac [New York Heart Association Class III or IV] or respiratory disease).
* Anticoagulants (other than LMWH or heparin in prophylactic doses to prevent deep vein thrombosis), direct thrombin inhibitors or thrombolytic therapy administered or completed within last week.
* Jehovah's Witnesses, or any other group of patients with ethical objections to receiving blood products.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Blood loss as calculated from change in haematocrit | 7 days

SECONDARY OUTCOMES:
Intra-operative blood loss | 1 day
Postoperative blood loss | postoperative 4 hours, 1 day, 2 days, 7days respectively
Hemoglobin levels | postoperative 4 hours, 1 day, 2 days, 7days respectively
drainage volume | postoperative 1 day, 2 days
Proportion of patients receiving transfusions | 7 days
Incidence of deep vein thrombosis postoperatively | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Yong Li, Principal Investigator — The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Locations (1):
- the First Affiliated Hospital of Guangzhou TCM University, Guangzhou, Guangdong, China